CLINICAL TRIAL: NCT07345143
Title: Artificial Intelligence in Education and Monitoring Women With Gestational Diabetes
Brief Title: Artificial Intelligence and Gestacional Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: JOSE FERNANDO VILELA-MARTIN (Other)
Responsible Party: Sponsor-Investigator, JOSE FERNANDO VILELA-MARTIN, MD, PHD, Hospital de Base
Organization: Hospital de Base (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78204024.6.0000.5415.
Record Dates: First submitted 2025-11-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-01

CONDITIONS: Gestational Diabetes; Macrosomia, Fetal
Keywords: artificial intelligence; gestacional diabetes; machine learning; glucose monitoria; glucose sensor
MeSH Terms: conditions — Diabetes, Gestational; Fetal Macrosomia | interventions — Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device group: Case group (AI model use) (Experimental): Case group - Device group. AI model to monitor glucose control and send education to treat women with gestacional diabetes in insulin treatment.
  Interventions: Other: monitoring model for women with gestacional diabetes using pharmacological therapy
- Control group (no use of AI model) (No Intervention): No device group: Control group - women with gestacional diabetes in insulin treatment under conventional treatment, without the AI model use.

INTERVENTIONS:
Other: monitoring model for women with gestacional diabetes using pharmacological therapy — Artificial Intelligence modell through WhatsApp® to remote monitoring gestacional diabetes in insulin treatment, focusing on disease education, glycemic control monitoring, and therapeutic interventions.
  Other Names: artificial intelligence for women with gestacional diabetes
  Arms: Device group: Case group (AI model use)

SUMMARY:
Artificial intelligence (AI) technology can assist medical teams in remote monitoring and continuing education of women with gestational diabetes (GDM), potentially improving adherence to interventions and impacting outcomes. An AI remote monitoring model called "monitoring model for women with GDM using pharmacological therapy," created by the ChamouDr technical team, will be analyzed focusing on disease education, glycemic control monitoring, and therapeutic interventions. Women diagnosed with GDM are invited to participate in the study and sign a free and informed consent form. The AI tool is installed on the pregnant woman's cell phone, who receives instructions to collect capillary blood glucose 6 times a day according to the protocol, at home, and report the results via WhatsApp to the study tool. Algorithm generated by the AI model based on self monitoring of blood glucose (SMBG) informs about diabetes control in the last week. The dashboard is accessible via a web browser, and signals: in green and red for patients with satisfactory and unsatisfactory control, respectively. Thus, the AI model optimizes the team's time in analyzing and treating patients appropriately in a simple, cost-effective, and accessible way.

DETAILED DESCRIPTION:
AI technology can assist medical teams in remote monitoring and continuing education of women with GDM. Objective: To analyze the results of using an AI model in remote monitoring and continuing education of women with GDM and pharmacological treatment, correlating them with clinical outcomes for the mother-fetus binomial. Methods: prospective, longitudinal, interventional clinical study approved by the local ethics committee. Patients signed a consent form to participate. An AI remote monitoring model called "monitoring model for women with GDM using pharmacological therapy," created by the ChamouDr technical team, will be analyzed focusing on disease education, glycemic control monitoring, and therapeutic interventions. The modell uses WhatsApp®, through a structured chatbot and AI resources, to communicate with the participant. Comparative analyses will be conducted between two groups of 100 pregnant women with GDM on insulin therapy, followed in the high-risk prenatal clinic of the Obstetrics Department of a tertiary hospital: case group using the AI model versus control group, composed of patients previously monitored under conventional in-person supervision, without the use of this technology. Algorithm generated by the AI model based on SMBG informs about diabetes control in the last week. The dashboard is accessible via a web browser, and signals: in green and red for patients with satisfactory and unsatisfactory control, respectively. Thus, the AI model optimizes the team's time in analyzing and treating patients appropriately in a simple, cost-effective, and accessible way.

ELIGIBILITY:
Inclusion Criteria:

* Gestacional diabetes women with gestational age of up to 28 weeks and 6 days
* Gestacional diabetes women who sign the free and informed consent form

Exclusion Criteria:

* Gestational age greater than 28 completed weeks at the first consultation
* Participants with overt DM (fasting glucose > 126 mg/dl or postprandial > 200 mg/dl)
* Unknown outcome.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only Women
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
fetal death | From the moment of randomization to delivery (until 40 weeks of pregnancy)
  Fetal death resulting from metabolic changes caused by gestational diabetes
Fetal birth weight | From the moment of randomization to delivery (until 40 weeks of pregnancy)
  Fetal weight at birth assessed using a precision scale.
neonatal hypoglycemia | From the moment of randomization to delivery (until 40 weeks of pregnancy), and Assessment of neonatal blood glucose levels from birth up to 48 hours post-birth.
  Neonatal hypoglycemia is the abnormal reduction of glucose in the newborn's blood to levels considered insufficient to meet the metabolic needs of the brain and other tissues. Plasma glucose parameters:
  < 40 mg/dL in the first 4 hours of life, < 45 mg/dL between 4 and 24 hours of life, After 24 hours, values < 50-60 mg/dL
glycemic control | From the moment of randomization to delivery (until 40 weeks of pregnancy)
  Glycemic control will be evaluated according to capillary glucose measurements that are taken 6 times a day: fasting, before and 1 hour after meals, following the target ranges of 70 to 95 mg/dL fasting; 70 ton 100 mg/dL pre-prandial; and 100 to 140 mg/dL post-prandial.

SECONDARY OUTCOMES:
admission of the newborn to the intensive care unit | From the moment of randomization to delivery (until 40 weeks of pregnancy), and from birth to 48 hours postpartum
  The need for the newborn to be admitted to an intensive care unit due to metabolic disorders associated with poor maternal glycemic control.
mother weight gain | From the moment of randomization to delivery (until 40 weeks of pregnancy).
  Maternal weight gain assessed during the gestational follow-up period up to delivery.
gestational age at delivery | From the moment of randomization to delivery (until 40 weeks of pregnancy).
  Gestational age at the time of natural childbirth or cesarean section in weeks
route of delivery | From the moment of randomization to delivery (until 40 weeks of pregnancy).
  Description of whether it was a natural birth or a cesarean section.
Blood pressure | From the moment of randomization to delivery (until 40 weeks of pregnancy).
  Evaluate if hypertension is present and assess blood pressure levels during pregnancy and up to delivery.

CONTACTS AND LOCATIONS:
Overall Officials: José F Vilela-Martin, MD, PhD, Principal Investigator — Hospital de Base; Vanessa V Goulart, MD, MSc, Principal Investigator — Hospital de Base, Sao Jose do Rio Preto, Sao Paulo, Brazil; Ligia C Junqueira, MD, Study Chair — Hospital de Base, Sao Jose do Rio Preto, Sao Paulo, Brazil; Amanda T Lotierzo, MD, Study Chair — Hospital de Base, Sao Jose do Rio Preto, Sao Paulo, Brazil; Carolina C Amorim, MD, Study Chair — Hospital de Base, Sao Jose do Rio Preto, Sao Paulo, Brazil; Maria Amalia BC Cançado, MD, Study Chair — Hospital de Base, Sao Jose do Rio Preto, Sao Paulo, Brazil; Leticia A Mantoani, student, Study Chair — Hospital de Base, Sao Jose do Rio Preto, Sao Paulo, Brazil; Rodrigo F Zancaner, Study Chair — Chamoudr company; Rafael Beolchi, Study Chair — Chamoudr company; Lucas F Queiroz, Study Chair — Chamoudr company; Luciana N Cosenso-Martin, MD, PhD, Study Chair — Hospital de Base, Sao Jose do Rio Preto, Sao Paulo, Brazil
Locations (1):
- Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dhombres F, Bonnard J, Bailly K, Maurice P, Papageorghiou AT, Jouannic JM. Contributions of Artificial Intelligence Reported in Obstetrics and Gynecology Journals: Systematic Review. J Med Internet Res. 2022 Apr 20;24(4):e35465. doi: 10.2196/35465. PMID 35297766
- [Background] Akazawa M, Hashimoto K. Artificial intelligence in gynecologic cancers: Current status and future challenges - A systematic review. Artif Intell Med. 2021 Oct;120:102164. doi: 10.1016/j.artmed.2021.102164. Epub 2021 Sep 3. PMID 34629152
- [Background] Grunebaum A, Chervenak J, Pollet SL, Katz A, Chervenak FA. The exciting potential for ChatGPT in obstetrics and gynecology. Am J Obstet Gynecol. 2023 Jun;228(6):696-705. doi: 10.1016/j.ajog.2023.03.009. Epub 2023 Mar 15. PMID 36924907
- [Background] Sweeting A, Wong J, Murphy HR, Ross GP. A Clinical Update on Gestational Diabetes Mellitus. Endocr Rev. 2022 Sep 26;43(5):763-793. doi: 10.1210/endrev/bnac003. PMID 35041752
- [Background] Ye W, Luo C, Huang J, Li C, Liu Z, Liu F. Gestational diabetes mellitus and adverse pregnancy outcomes: systematic review and meta-analysis. BMJ. 2022 May 25;377:e067946. doi: 10.1136/bmj-2021-067946. PMID 35613728
- [Background] Mistry SK, Das Gupta R, Alam S, Kaur K, Shamim AA, Puthussery S. Gestational diabetes mellitus (GDM) and adverse pregnancy outcome in South Asia: A systematic review. Endocrinol Diabetes Metab. 2021 Oct;4(4):e00285. doi: 10.1002/edm2.285. Epub 2021 Jul 3. PMID 34505412
- [Background] Ugwudike B, Kwok M. Update on gestational diabetes and adverse pregnancy outcomes. Curr Opin Obstet Gynecol. 2023 Oct 1;35(5):453-459. doi: 10.1097/GCO.0000000000000901. Epub 2023 Aug 9. PMID 37560815
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375